

# Non-Interventional Study (NIS) Protocol

| Document Number: | c41847952-01 |
|---|---|
| BI Study Number: | 1199-0526 |
| BI Investigational Product(s): | Nintedanib |
| Title: | Assessment of the Dose Reduction and Discontinuation associated with Anti-Fibrotic Medications in Patients with Idiopathic Pulmonary Fibrosis |
| Brief lay title: | Dose Reduction and Discontinuation with Anti-Fibrotic Medications |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | Not applicable |
| PASS: | Pending |
| EU PAS register<br>number: | Pending |
| Active substance: | NA |
| Medicinal product: | Nintedanib (Ofev) and Pirfenidone (Esbriet) |
| Product reference: | NA NA |
| Procedure number: | Not applicable |
| Marketing authorisation holder(s): | NA NA |
| Joint PASS: | Not applicable |
| Research question and objectives: | Primary aim - To assess average daily dose, and dose reduction/interruption patterns in nintedanib and pirfenidone initiators separately at 6- and 12- months post-initiation. |
| | Secondary aim - To assess drug discontinuation patterns in nintedanib and pirfenidone initiators separately at 6- and 12-months post-initiation. |

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Country(-ies) of study: | United States |
|--------------------------------------|----------------|
| Authors: | |
| Marketing authorisation holder(s): | Not applicable |
| Date: | 24 MAR 2023 |
| Proprietary confidential information | |

© 2023 Boehringer Ingelheim Group of companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. TABLE OF CONTENTS

| TITL | E PAG | E 1 |
|---|---|---|
| 1. | TABL | E OF CONTENTS |
| 2. | LIST ( | OF ABBREVIATIONS5 |
| 3. | RESPO | ONSIBLE PARTIES6 |
| 4. | ABSTI | RACT |
| 5. | AMEN | IDMENTS AND UPDATES10 |
| 6. | MILES | STONES11 |
| 7. | RATIO | DNALE AND BACKGROUND12 |
| 8. | RESEA | ARCH QUESTION AND OBJECTIVES14 |
| 9. | RESEA | ARCH METHODS15 |
| 9.1 | STU | JDY DESIGN15 |
| 9.2 | SET | TTING 16 |
| 9 | .2.1 | Study sites |
| 9 | .2.2 | Study population |
| 9 | .2.3 | Study visits |
| 9 | .2.4 | Study discontinuation |
| 9.3 | VA | RIABLES |
| 9 | .3.1 | Exposures |
| 9 | .3.2 | Outcomes |
| | 9.3.2.1 | - |
| | 9.3.2.2 | |
| _ | .3.3 | Covariates |
| 9.4 | | TA SOURCES |
| | | JDY SIZE 23 |
| 9.6 | | TA MANAGEMENT |
| 9.7 | | TA ANALYSIS |
| | .7.1 | Main analysis |
| | .7.2 | Post-hoc analysis |
| 9.8<br>9.9 | | ALITY CONTROL |
| | | HER ASPECTS25 |
| | | [11] (IX / XX ) [1 X / 1 X X X X X X X X X |

| NIS Protocol | |
|---|---|
| Study number: 1199-0526 | Document number: c41847952-01 |
| Proprietary confidential information © 2023 Boehringer Ingelheim International | d GmbH or one or more of its affiliated companies |
| 9.10.1 Data quality assurance | 26 |
| 9.10.2 Study records | 26 |
| 10. PROTECTION OF HUMAN SUBJECTS | 27 |
| 10.1 STUDY APPROVAL, PATIENT INFORMAT CONSENT | |
| 10.2 STATEMENT OF CONFIDENTIALITY | 27 |
| 11. MANAGEMENT AND REPORTING OF ADVEREACTIONS | |
| 11.1 ADVERSE EVENT AND SERIOUS ADVER REPORTING | |
| 12. PLANS FOR DISSEMINATING AND COMMU | |
| 13. REFERENCES | 30 |
| 13.1 PUBLISHED REFERENCES | 30 |
| ANNEXES | 32 |
| ANNEX 1. LIST OF STAND-ALONE DOCUMENT | S32 |
| ANNEX 2. ENCEPP CHECKLIST FOR STUDY PRO | OTOCOLS 33 |
| ANNEX 3. ADDITIONAL INFORMATION | 34 |
| ANNEY A DEVIEWEDS AND ADDROVAL SIGNA | TURES 35 |

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event

AESI Adverse Event of Special interest

CA Competent Authority
CCDS Company Core Data Sheet

CI Confidence Interval
CML Local Clinical Monitor
CRA Clinical Research Associate

CRF Case Report Form

CTCAE Common Terminology Criteria for Adverse Events

CTP Clinical Trial Protocol

eCRF Electronic Case Report Form

ENCePP European Network of Centres for Pharmacoepidemiology and

Pharmacovigilance

FDA Food and Drug Administration

GCP Good Clinical Practice

GEP Good Epidemiological Practice

GPP Good Pharmacoepidemiology Practice GVP Good Pharmacovigilance Practices

IB Investigator's Brochure

IEC Independent Ethics Committee
IRB Institutional Review Board
MAH Marketing Authorization Holder

MedDRA Medical Dictionary for Regulatory Activities

NIS Non-Interventional Study

PASS Post-Authorization Safety Study

SAE Serious Adverse Event USD United States Dollar

NIS Protocol

Study number: 1199-0526
Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 3. RESPONSIBLE PARTIES

| BI NIS | İ |
|------------|---|
| BI NIS co- | |

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. ABSTRACT

| Name of company | : | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: Nintedanib (Ofev) and Pirfenidone (Esbriet) | | | |
| Name of active ing<br>Nintedanib (Ofev) a<br>Pirfenidone (Esbrie | and | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 24 MAR 2023 | 1199-0526 | | |
| Title of study: | Assessment of the Dose Reduction/Interruption and Discontinuation with Nintedanib and Pirfenidone Initiators in Patients with Idiopathic Pulmonary Fibrosis | | |
| Rationale and background: | Antifibrotics have demonstrated an ability to slow IPF progression, if taken according to the recommended dosing and taken continuously, in both clinical trials and real-world evidence. Previous real-world studies have compared persistence/discontinuation patterns for nintedanib and pirfenidone and found similar persistence patterns for both drugs. However, these studies have failed to consider the differential dosing regimens between these two drugs and corresponding incidence of dose reduction/interruption. This study will assess both dose reduction/interruption and discontinuation patterns for nintedanib and pirfenidone among patients with IPF. | | |
| Research question and objectives: | <ol> <li>Primary aim - To assess average daily dose, and corresponding dose reduction/interruption patterns in nintedanib and pirfenidone initiators separately at 6- and 12-months post-initiation.</li> <li>Secondary aim - To assess drug discontinuation patterns in nintedanib and pirfenidone initiators separately at 6- and 12-months post-initiation.</li> </ol> | | |
| Study design: | This is a non-interventional, retrospective cohort study with existing data. | | |

NIS Protocol 

| Name of company | :<br>: | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: Nintedanib (Ofev) and Pirfenidone (Esbriet) | | | |
| Name of active ing<br>Nintedanib (Ofev) a<br>Pirfenidone (Esbrie | and | | |
| Protocol date: 24 MAR 2023 | Study<br>number:<br>1199-0526 | Version/Revision: | Version/Revision date: |
| Population: | The study sample will consist of patients with IPF who initiated either nintedanib or pirfenidone between October 2014 to September 2021. The study will use data from the Optum Research Database (ORD), a claims database containing approximately 14 million commercial enrollees and 4 million Medicare-advantage enrollees | | |
| Variables: | The main outcome of our study will be incidence of dose reduction/interruption, calculated separately for nintedanib and pirfenidone. For each patient, average daily dose will be calculated in pre-specified time-periods (for example – the first 6 months, the first 12 months, and the average daily dose calculated separately in each month since drug initiation). Incidence of dose reduction/interruption will be defined as average daily dose not following the prescribing information. | | |
| | As a secondary outcome, we will also assess drug discontinuation during first 6 and 12 months separately for pirfenidone and nintedanib and will be defined as a gap of at least 60 days in filling of prescription (a gap of 60 days after the prescription date + days of supply for the current prescription). | | |
| Data sources: | We will use administrative health insurance claims data from the Optum Research Database (ORD) for the period of October 1, 2013 through end of data availability (currently September 30, 2022). This database was chosen as it includes claims of Medicare Advantage and commercially enrolled beneficiaries. | | |
| Study size: | As this is a descriptive study, no formal calculation of sample size was performed. In a preliminary feasibility analysis using Optum data to examine sample size, we have found that 1,979 patients newly | | |

NIS Protocol 

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished a product: Nintedanib (Ofev) : Pirfenidone (Esbrie | and | | |
| Name of active ing<br>Nintedanib (Ofev) :<br>Pirfenidone (Esbrie | and | | |
| Protocol date: | Study number: | Version/Revision: | Version/Revision date: |
| 24 MAR 2023 | 1199-0526 | | |
| | initiated pirfenidone, and 2,559 patients who initiated nintedanib between 10/2014 to 12/2020. As such, this study is expected to have a sufficient sample. | | |
| Data analysis: | Average daily dose during first 6 months and 12 months after drug initiation will be reported as means with standard deviations (SD), and median with interquartile range. Six months and 12-months daily dose categories will be presented as frequencies with percentages. Incidence of dose reduction/interruption will be reported by month of occurrence (using month 2 and onwards) and reported as frequencies with percentages. Drug discontinuation will be reported as frequencies with percentages, and time to drug discontinuation will be reported in months (mean (SD)). As this is a descriptive study, there will be no multivariable adjustment and/or direct comparison of outcomes between the pirfenidone and nintedanib cohort. | | |
| Milestones: | The analytic database is expected to be constructed by April 20, 2023, and data analyses are expected to be completed by May 15, 2023. A draft report of the findings from this study is expected to be available for review by June 15, 2023 and completed by August 30, 2023. | | |

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. AMENDMENTS AND UPDATES

None.

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6. MILESTONES

| Milestone | Planned Date |
|------------------------------|--------------|
| First draft of summary | 09/26/2022 |
| AET summary review | 10/17/2022 |
| NPCC summary review | 12/02/2022 |
| Study protocol first draft | 01/31/2023 |
| NIS disclosure review | 02/28/2023 |
| Analytical database creation | 04/20/2023 |
| Descriptive results | 05/15/2023 |
| Final report first draft | 06/15/2023 |

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. RATIONALE AND BACKGROUND

Idiopathic pulmonary fibrosis (IPF) is a life-threatening rare disease characterized by decline in lung function due to progression of fibrosis in the interstitium of the lung [1]. In patients with IPF, a decline in forced vital capacity (FVC) is an important indicator of mortality [6]. The median survival of non-treated IPF patients is approximately 3 years from diagnosis [2].

Before anti-fibrotic medications became available in the US, IPF treatment mainly consisted of therapeutics that were found not to be of benefit (or even harmful), and a mainstay of care focused on symptom relief and included palliative care [3]. In October 2014, two anti-fibrotic medications, nintedanib and pirfenidone, were approved by the U.S. Food and Drug Administration (FDA) for the treatment of IPF [4, 5], which transformed the treatment of this disease. Both medications were found to reduce the rate of decline in FVC compared to placebo in phase III clinical trials [7, 8].

From the perspective of treatment, the approvals of antifibrotics for IPF were significant breakthroughs. Antifibrotics have demonstrated an ability to slow IPF progression, if taken according to the recommended dosing in the prescriber information and taken continuously, in both clinical trials [7, 8] and real-world evidence [9]. Previous real-world studies have compared persistence/ discontinuation patterns for pirfenidone and nintedanib and found similar persistence patterns for both drugs [10, 11]. However, these studies have failed to consider the differential dosing regimens between these two drugs and corresponding incidence of dose reduction and/or temporary dose interruption. Hence, this study will assess both dose reduction and/or temporary dose interruption and discontinuation patterns for pirfenidone and nintedanib among patients with IPF.

In this study, we will investigate the incidence of dose reduction/interruption beyond the label recommendations (defined as a dose not following the prescriber information (PI), which corresponds to a daily dose of 2165 mg (90% of full dose, which is 2403 mg) for pirfenidone [12, 13] or less than a daily dose of 200 mg for nintedanib (66.67% of full dose, which is 300 mg) [14]) from 10/01/2014 to 09/30/2022 using real-world data. The definition of incidence of dose reduction, which is differential for nintedanib and pirfenidone is because of –

- 1) In the US, the prescriber information (PI) and/or label for pirfenidone does not indicate any particular dose reduction recommended as per Food & Drug Administration (FDA). For nintedanib, reducing dose from 150 mg to 100 mg BID is part of the PI.
- 2) The post-hoc analysis of clinical trials showed similar slope of FVC decline for patients who reduced the dose to 100 mg BID for nintedanib, but for pirfenidone, the slope of FVC decline was steeper for patients who reduced the dose, potentially indicating that reduced dose might lead to lower benefit on FVC decline (see figures below) [12, 15]

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



The current study may be able to demonstrate to decision makers the differential complexities in dosing regimen for pirfenidone vs. nintedanib and may reveal that IPF patients may not be receiving the full benefit of pirfenidone due to possible sub-optimal dosing, even when the patient has not discontinued the drug.

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. RESEARCH QUESTION AND OBJECTIVES

The overarching aim of our study is to assess the incidence of dose reduction and discontinuations separately for pirfenidone and nintedanib. Specific objectives are:

Primary aim - To assess average daily dose, and corresponding dose reduction/interruption patterns in pirfenidone initiators and nintedanib initiators separately at 6- and 12- months post-initiation.

Secondary aim - To assess drug discontinuation patterns in pirfenidone initiators and nintedanib initiators separately at 6- and 12-months post-initiation.

001-MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This study will be a retrospective cohort, descriptive study of patients with idiopathic pulmonary fibrosis (IPF). Patients with IPF who initiated either pirfenidone or nintedanib between October 2014 to September 2021 will be identified. The study will use data from the Optum Research Database (ORD), a claims database containing approximately 14 million commercial enrollees and 4 million Medicare-advantage enrollees. The date of the first prescription of either pirfenidone or nintedanib will be assigned as index date. Two separate cohorts will be created - 1) pirfenidone initiators, and 2) nintedanib initiators, and all outcomes will be assessed in the 12 months post-index period. A 12-month time-period prior to the index date will be used as the baseline period for determining the characteristics of patients in both cohorts. To allow for a 12-months baseline and follow-up periods for all patients, the span of data will be from 10/01/2013 to 09/30/2022. (Figure 1)



Figure 1 Study Design Schematic

The main outcome of our study will be incidence of dose reduction/interruption, calculated separately for pirfenidone and nintedanib. For each patient, average daily dose will be calculated in pre-specified time-periods (for example – the first 6 months, the first 12 months, and the average daily dose calculated separately in each month since drug initiation) (more details in section 2.6). Incidence of dose reduction/interruption will be defined as average daily dose not following the prescribing information (PI). According to the PI, the daily dose of pirfenidone is 2403 mg [13], hence the study will consider average daily dose less than 2165 mg (90% of PI dose) as dose reduction for pirfenidone [12]. For nintedanib, the daily dose allowed under prescriber information is 200 mg [14], hence less than 200 mg will be considered a dose reduction for nintedanib patients. As a secondary outcome, we will also assess drug discontinuation during first 6 and 12 months separately for pirfenidone and nintedanib and will be defined as a gap of at least 60 days in filling of prescription (a gap of 60 days after the prescription date + days of supply for the current prescription). In a sensitivity analysis, we will explore 30- and 90- days gap as a definition for drug discontinuation. As this is a descriptive study, assessment of the dose reduction and discontinuation for both drugs will be considered separately, and only descriptively, without any direct comparison between the two cohorts.

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2 SETTING

#### 9.2.1 Study sites

We will use administrative health insurance claims data from the Optum Research Database (ORD) for the period of October 1, 2013 through end of data availability (currently September 30, 2021). The ORD contains enrollment information, as well as fully-adjudicated medical claims and pharmacy claims for commercial enrollees and MAPD beneficiaries. In 2018, the ORD included 14.3 million commercial enrollees with medical and pharmacy benefits and 4.3 million beneficiaries with Medicare Part C (commonly referred to as the Medicare Advantage program). Medicare Advantage beneficiaries choose to receive all of their health care services through a provider organization in lieu of Medicare Part A/B coverage (commonly referred to as Medicare Fee for Service). These plans are referred to as MAPD when combined with Medicare Part D coverage. The average enrollment duration was 31.4 and 37.3 months for commercial enrollees and MAPD enrollees, respectively. Underlying information is geographically diverse across the United States and enrollees are fairly representative of the U.S. population. Medicare beneficiaries retain a single identifier within the system and can be tracked as they change plans, or as they disenroll and reenroll over time.

Claims for pharmacy services are typically submitted electronically by the pharmacy at the time prescriptions are filled. The claims history is a profile of all outpatient prescription pharmacy services provided and covered by the health plan. Pharmacy claims data include drug name, dosage form, drug strength, fill date, days of supply, financial information, and de-identified patient and prescriber codes, allowing for longitudinal tracking of medication refill patterns and changes in medications. Pharmacy claims are typically added to the research database within six weeks of dispensing.

Medical claims or encounter data are collected from all available health care sites (inpatient hospital, outpatient hospital, emergency department, physician's office, surgery center, etc.) for virtually all types of provided services, including specialty, preventive and office-based treatments. Medical claims and coding conform to insurance industry standards. Claims for ambulatory services submitted by individual providers, such as physicians, use the Health Care Financing Administration (HCFA)-1500 or Centers for Medicare and Medicaid Services (CMS)-1500 formats. Claims for facility services submitted by institutions, e.g., hospitals, use the Uniform Billing (UB)-82, UB-92, UB-04, or CMS-1450 formats. Medical claims include: multiple diagnosis codes recorded with the International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) and International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) diagnosis codes; procedures recorded with ICD-9-CM and ICD-10-CM procedure codes, Current Procedural Terminology (CPT), or Health care Common Procedure Coding System (HCPCS) codes; site of service codes; provider specialty codes; revenue codes (for facilities); paid amounts; and other information. Typically, facility claims do not include medications dispensed in hospital. Approximately six months following the delivery of services is required for complete adjudication of medical data.

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2.2 Study population

For the primary study objective, patients included in the cohort need to meet the following criteria:

- Presence of at least one pirfenidone or nintedanib prescription during the identification period (the date of first prescription for pirfenidone/nintedanib is the index date)
- Evidence of IPF: patient with at least one inpatient or two outpatient claims (>14 days apart) with a diagnosis code for IPF (ICD-10-CM: J84.112; ICD-9-CM: 516.31) during the study period (10/01/2013 to 09/30/2022)
- At least 18 years old at the index date
- Have at least 12 months of continuous enrollment in the health plan during pre-index period, and at least 6 months of continuous enrollment in post-index period (for 12-months analysis, patients would be required to have 12 months post-index continuous enrollment)

Exclusion criteria include the following:

- Any history of lung transplant during the 12-months pre-index/baseline period
- Any claims for a skilled nursing facility, a long-term care facility or hospice care during the 12-month pre-index period
- Evidence (≥2 ICD-9-CM or ICD-10-CM diagnostic codes on different dates) of non-IPF chronic fibrosis ILD or connective tissue diseases during the 12-months pre-index period. The following conditions will be excluded: autoimmune, or connective tissue diseases (i.e., rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), dermatopolymyositis, systemic sclerosis, Sjogren's syndrome, and mixed connective tissue disease (CTD)), sarcoidosis, and hypersensitivity pneumonitis).
- Missing demographic information (i.e., age or sex)

#### 9.2.3 Study visits

Not applicable

#### 9.2.4 Study discontinuation

Not applicable.

#### 9.3 VARIABLES

#### 9.3.1 Exposures

There is no primary exposure in this study, as this is a descriptive study evaluating dose reduction/interruption, and drug discontinuation in pirfenidone and nintedanib initiators, separately. There is no direct comparison between the two cohorts (more details in <u>Section</u> 9.7)

NIS Protocol 

**Study number: 1199-0526 Document number: c41847952-01** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3.2 Outcomes

#### 9.3.2.1 Primary outcome

The main outcome measure of our study is the incidence of dose reduction/interruption, calculated separately for each drug. For calculating the primary outcome, we will first need to calculate the average daily dose of pirfenidone and nintedanib after drug initiation (post-index period). Specific details of calculations are —

Average daily dose

Average daily dose for each patient will be calculated by taking the average of total drug intake (tablet strength \* number of doses) during the time between index date to the date of drug discontinuation

```
Average \ Daily \ Dose \\ = \frac{\sum_{0}^{n}(Tablet \ Strength*number \ of \ tablets \ in \ a \ Rx \ fill)}{Time \ of \ follow - up \{(Date \ of \ discontinuation) - Index \ Date\}} Where n = number of fills a patient has received for pirfenidone/nintedanib
```

- We will calculate average daily dose of pirfenidone and nintedanib separately for each month in post-index period (month 1 to 12) and will also calculate for cumulative periods of 6 months and 12 months. For all calculations, censoring events will be taken into account, with patient censored at the date of drug discontinuation, or end of 12 months.
- Six and twelve months average daily dose categories For the average daily dose calculations in cumulative periods, we will be dividing the patients in following 4 categories
  - 1) Dose strength less than 50%
  - 2) Dose strength between 51% to 66%
  - 3) Dose strength between 67% to 90%
  - 4) Dose strength above 90%

#### Incidence of Dose Reduction and/or temporary dose interruption

Once average daily dose is calculated for each month post-index (month 1 to 12), incidence of dose reduction/interruption will be calculated as presence of average daily dose  $\leq 90\%$  dose strength (for pirfenidone) or  $\leq 66.67\%$  dose strength (for nintedanib), as per the PI [12 – 14]. Patients will be required to have the dose reduction for at least for 60 days, to make sure that the dose reduction is not temporary.

In a sensitivity analysis, we will also evaluate temporary dose reductions, i.e., dose reduced to below the above defined dose strength only for 1 month.

In the primary analysis, patients who reduce their dose in the prior months will be allowed to discontinue the drug in future months (For example, in primary analysis, a patient can reduce their index drug dose in month 2 (i.e. dose below label recommendation for the whole month 2 and 3), and then can discontinue the drug in month 4 (or beyond). We will also evaluate the incidence of dose reduction in patients who never discontinue the index drug.

NIS Protocol 

**Study number: 1199-0526 Document number: c41847952-01** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 9.3.2.2 Secondary outcomes

We will assess drug discontinuation as a secondary outcome. Pirfenidone or nintedanib discontinuation will be defined as presence of sixty or more days gap in refilling a prescription of the drug (sixty days gap counted from the date of last fill plus the days of supply for the fill). The date of last fill plus the days of supply for the fill (typically 30 days) will be designated as date of discontinuation, and time to discontinuation will be calculated as time between date of discontinuation and index date (only for patients who discontinue the drug). We will calculate the percentage of patients who discontinue each drug in first 6- and 12-months post-index period. As a sensitivity analysis, we will calculate drug discontinuation using 30 days and 90 days as allowed gap between the scripts (vs. 60 days)

We will also assess how many patients initiate either of the antifibrotic drugs (including the same drug the patient has discontinued) during the follow-up time post discontinuation of their index drug. We will separately assess initiation of the index drug vs. initiation of the other antifibrotic agent.

#### 9.3.3 Covariates

| Variable | Description |
|---|---|
| Demographic and socioeconomic characteristics | |
| Age | Age as of index date in whole years will be calculated based on the difference between the patient's birth date and index date. |
| Women | Women will be a binary indicator for whether the beneficiary was woman as indicated on the enrollment record covering the index date. |
| Census region | Census region will be a categorical variable defined by categorizing the beneficiary's state of residence into Census regions (Northeast, South, Midwest, West) from the enrollment record covering the index date |
| Index year | Index year will be a categorical variable defined as the year of the index date and will take the values 2014, 2015 2016, 2017, 2018, 2019, 2020 or 2021. |
| Clinical characteristics | |
| Charlson Comorbidity Index (CCI) | Charlson Comorbidity Index (CCI) during pre-<br>index period: A CCI score will be calculated for<br>each patient using diagnosis codes on medical<br>claims during the pre-index period. The CCI was<br>developed in 1987 based on 1-year mortality data |

NIS Protocol 

| Variable | Description |
|---|---|
| | from internal medicine patients, and encompasses 19 medical conditions weighted 1–6 with total scores ranging from 0–37 (Charlson ME 1987). For this study, CCI adapted for use with both ICD-9-CM and ICD-10 codes will be used (Quan H 2005). The CCI will be reported as both a continuous measure and a categorical measure (0=low, 1-2=medium, or ≥3=high). |
| Pulmonary hypertension | A binary indicator for whether the beneficiary had<br>a diagnosis code for pulmonary hypertension on at<br>least one inpatient, or outpatient claim that<br>occurred during the baseline period |
| Gastroesophageal reflux disease (GERD) | A binary indicator for whether the beneficiary had a diagnosis code for gastroesophageal reflux disease on at least one inpatient, or outpatient claim that occurred during the baseline period |
| Asthma | A binary indicator for whether the beneficiary had<br>a diagnosis code for asthma on at least one<br>inpatient, or outpatient claim that occurred during<br>the baseline period |
| Sleep apnea | A binary indicator for whether the beneficiary had<br>a diagnosis code for obstructive sleep apnea on at<br>least one inpatient, or outpatient claim that<br>occurred during the baseline period |
| Lung biopsy | A binary indicator for whether the beneficiary had<br>a diagnosis or procedure code for a lung biopsy on<br>at least one inpatient, or outpatient claim that<br>occurred during the baseline period |
| HRCT scan | A binary indicator for whether the beneficiary had a procedure code for a high-resolution computerized tomography scan on at least one inpatient, or outpatient claim that occurred during the baseline period |
| Oxygen | A binary indicator for whether the beneficiary had<br>a diagnosis, procedure revenue center code for<br>oxygen therapy or supplemental oxygen on at<br>least one inpatient, outpatient, skilled nursing<br>facility, home health or durable medical |

NIS Protocol 

| Variable Description | |
|---|---|
| | equipment claim that occurred during the baseline period |
| Pulmonary rehabilitation | A binary indicator for whether the beneficiary had a procedure or revenue center code for pulmonary rehabilitation services on at least one inpatient, outpatient, skilled nursing facility, home health or durable medical equipment claim that occurred during the baseline period |
| Ventilator use | A binary indicator for whether the beneficiary had<br>a diagnosis or procedure code for ventilator use on<br>at least one inpatient, or outpatient claim that<br>occurred during the baseline period |
| COPD | A binary indicator for whether the beneficiary had<br>a diagnosis code for chronic obstructive<br>pulmonary disease on at least one inpatient, or<br>outpatient claim that occurred during the baseline<br>period |
| Нурохіа | A binary indicator for whether the beneficiary had<br>a diagnosis code for hypoxia on at least one<br>inpatient, or outpatient claim that occurred during<br>the baseline period |
| Pharmacy use and spending | |
| Medication count | The count of the number of unique outpatient prescription medications for which beneficiary has pharmacy claims during the baseline period |
| Total pharmacy spending | A continuous, non-negative variable representing<br>the total amount paid by all parties for outpatient<br>prescription medications as reported in pharmacy<br>claims during the baseline period. |
| OOP pharmacy spending | A continuous, non-negative variable representing the total amount paid out-of-pocket by the beneficiary for outpatient prescription medications as reported in pharmacy claims during the baseline period. |
| Inpatient hospitalization use and spending | |
| Any inpatient stay | A binary indicator for whether a beneficiary had at least one inpatient hospitalization for any cause during the baseline period. |

NIS Protocol 

| Variable | Description |
|---|---|
| Inpatient stay count | A count of the number of inpatient hospitalizations for any cause a beneficiary had during the baseline period. |
| Inpatient length of stay | A count of the number of days (length of stay) a beneficiary was hospitalized in an inpatient facility during the baseline period. Length of stay for each inpatient hospitalization claim will be calculated as the arithmetic difference between each claim's from and through dates. |
| Total inpatient spending | A continuous, non-negative variable representing<br>the total amount paid by all parties for all inpatient<br>hospitalizations (for any cause) as reported in<br>inpatient facility claims during the baseline<br>period. |
| Outpatient facility use and spending | |
| Any outpatient visit | A binary indicator for whether a beneficiary had at least one claim for services provided by an outpatient facility for any cause during the baseline period. |
| Outpatient visit count | A count of the number of unique dates with an outpatient facility for any cause claim a beneficiary had during the baseline period. |
| Total outpatient spending | A continuous, non-negative variable representing the total amount paid by all parties for outpatient facility claims during the baseline period. |
| Medical spending | |
| Total Medical spending | A continuous, non-negative variable representing<br>the total amount paid by all parties all medical<br>claims during the baseline period, calculated as<br>the sum of the allowed amounts on each claim. |
| OOP Part B spending | A continuous, non-negative variable representing the total amount paid out-of-pocket by the beneficiary for all medical claims during the baseline period. |
| Total spending | |
| Total spending | A continuous non-negative variable representing the total amount paid by all parties for all medical |

NIS Protocol 

**Study number: 1199-0526 Document number: c41847952-01** 

| Proprietary confidential information © 2023 | Boehringer Ingelheim International | I GmbH or one or more of its affiliated companies |
|---|---|---|

| Variable | Description |
|---|---|
| | and pharmacy claims during the baseline period<br>and will be calculated as the sum of total<br>pharmacy and total medical spending. |
| Other use | |
| Any ED visit | A binary indicator for whether a beneficiary had at least one emergency department visit during the baseline visit. |
| ED visit count | A count of the number of unique dates with an emergency department visit that a beneficiary had during the baseline period. |
| Any pulmonology visit | A binary indicator for whether a beneficiary was treated by a specialist in pulmonary disease during the baseline period. Treatment by a pulmonologist will be identified by the presence of a pulmonary specialty code in inpatient, or outpatient claims. |
| Pulmonology visit count | A count of the number of unique dates with treatment by a specialist in pulmonary disease that a beneficiary had during the baseline period. |

#### 9.4 DATA SOURCES

As described above in <u>Section 9.2.1</u>, We will use administrative health insurance claims data from the Optum Research Database (ORD) for the period of October 1, 2013 through end of data availability (September 30, 2022). The ORD contains enrollment information, as well as fully-adjudicated medical claims and pharmacy claims for commercial enrollees and MAPD beneficiaries. In 2018, the ORD included 14.3 million commercial enrollees with medical and pharmacy benefits and 4.3 million beneficiaries with Medicare Part C (commonly referred to as the Medicare Advantage program).

#### 9.5 STUDY SIZE

As this is a descriptive study, no formal calculation of sample size was performed. In a preliminary feasibility analysis using Optum data to examine sample size, we have found that 1,979 patients newly initiated pirfenidone, and 2,559 patients who initiated nintedanib between 10/2014 to 12/2020. As such, this study is expected to have a sufficient sample.

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.6 DATA MANAGEMENT

Data cleaning and analysis will be executed by US HEOR group. Paper printouts of the data are not required and will not be produced. Study documents, including synopsis, protocol, final results, and publications, will be archived on the BIRDS (Boehringer Ingelheim Regulatory Documents for Submission).

#### 9.7 DATA ANALYSIS

#### 9.7.1 Main analysis

Baseline characteristics for the pirfenidone and nintedanib cohorts will be reported as frequencies with percentages for categorical data, and means with standard deviations (SD), and median with interquartile range will be reported for continuous variables. We will compare the baseline characteristics using Student's T-test or Wilcoxon rank-sum test for continuous variable, and chi-square test for categorical variable

Average daily dose during first 6 months and 12 months after drug initiation will be reported as means with standard deviations (SD), and median with interquartile range. Six months and 12-months daily dose categories will be presented as frequencies with percentages. Incidence of dose reduction will be reported by month of occurrence (using month 2 and onwards) and reported as frequencies with percentages. Time to drug dose reduction will be reported in months (mean (SD)). Drug discontinuation will be reported as frequencies with percentages, and time to drug discontinuation will be reported in months (mean (SD)). As this is a descriptive study, there will be no multivariable adjustment and/or direct comparison of outcomes between the pirfenidone and nintedanib cohort.

### 9.7.2 Post-hoc analysis

As this study is a descriptive analysis, no adjustments or direct comparison between pirfenidone and nintedanib cohort is proposed a-priori. If significant differences in the baseline characteristics between the pirfenidone and nintedanib cohorts are observed, we propose to conduct propensity score matching (PSM) to balance the baseline characteristics between the two cohort. Specifically, pirfenidone initiators will be matched to nintedanib initiators using the technique of nearest neighbor match on an estimated propensity score (caliper width of ±0.001 unit). The propensity score for this analysis will be obtained from a logistic regression model using pre-index measures to predict the probability of being in the pirfenidone initiator cohort. Pre-index measures which will be included are demographic (age, sex, census region, index year), clinical (CCI, pulmonary hypertension, COPD, asthma, GERD, HRCT scan, oxygen use, and ventilator use), and healthcare utilization measures (total pharmacy spend, total medical spend, number of pulmonology visits)

We will compare differences in baseline characteristics between the pirfenidone and nintedanib cohorts before and after propensity score matching. The success of the propensity score-matching to reduce confounding will be assessed by evaluating the standardized differences in the covariates between the study groups after matching. For each covariate, the standardized difference percent (di) will be calculated as:  $di = 100 * (xi - xni) / \sqrt{(s2i + xni)}$ 

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

s2ni}/2) where xi and xni are the sample means of the ith covariate in the pirfenidone and nintedanib cohorts, respectively, and s2i and s2ni are the corresponding sample variances. A standardized difference of <10% is considered an acceptable level of difference (or supports the assumption of balance) between the comparison groups.

We will reassess the primary and secondary outcomes in the matched cohorts (see <u>Section</u> 9.7.1 for more details)

#### 9.8 QUALITY CONTROL

The following quality assurance and quality control measures will be applied to all programming that executes data extraction and transformation by US HEOR team:

- Check program logs for notes, warning messages, and errors
- Check derived data values against source data for a patient sample to ensure correct derivation
- Verify that variables needed to support tables/listings/figures/ are found in the derived data set
- Check that data fields are not truncated
- Check data points for values outside expected ranges, where appropriate
- Check that data are rounded correctly and in accordance to the analysis plan
- Check that abbreviations, range categories, and subgroups conform to the analysis plan
- Ensure the consistency of sample counts across relevant tables/listings/figures
- Check formats consistent with the analysis plan
- Ensure no typos, misspellings, or false values
- Check that summary statistics are correct; check at least one category in each summary table against the data listings
- Check that data are in accordance with the Data Plan
- Check that subgroups conform to the Data Plan
- Ensure there are no duplicate observations

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

Several potential limitations of this study are discussed below:

- This study is based on healthcare claims data, daily dose calculations derived from monthly pharmacy fills may not represent the actual daily intake of the patient
- We could not ascertain reasons for discontinuations and/or dose reduction in this study, as adverse events may not be reliably captured in the claims database, and also the reasons for drug discontinuation are not captured in the claims database
- We will not be able to distinguish between dose reduction vs. temporary dose interruption for a patient, as the main outcome is based on calculation of daily dose based on pharmacy claims
- Due to lack of availability of laboratory data and clinical information (for example FVC% at baseline), severity of IPF, and results of the laboratory tests will not be

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

observed. The severity of IPF may influence the initiation, discontinuation, and dose-reduction of an anti-fibrotic agents

• This study cannot be generalized to the entire U.S. population. ORD only covers patients with commercial insurance or Medicare Advantage plan. The findings of this study may not be applicable for patients with public insurance such as Medicare Fee-For-Service or without insurance.

### 9.10 OTHER ASPECTS

## 9.10.1 Data quality assurance

See Section 9.8

## 9.10.2 Study records

Not applicable.

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10. PROTECTION OF HUMAN SUBJECTS

Not applicable.

# 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

IRB exemption has been granted to this study.

#### 10.2 STATEMENT OF CONFIDENTIALITY

IRB exemption has been granted to this study.

001-MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

Given the information available within the Optum claims database for this study, extraction on adverse events data will not be conducted and only data related to the study objectives will be extracted. Therefore, information about individual adverse events will not be available. Only data on aggregate-level medication use will be analyzed.

# 11.1 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

Not applicable based on secondary use of data without any potential that any employee of BI will access individually identifiable patient data.

001-MCS-90-118\_RD-23 (1.0) / Saved on: 25 Nov 2019

NIS Protocol 

**Study number: 1199-0526 Document number: c41847952-01** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The results of this study will be considered for dissemination in the form of scientific publications (e.g., an abstract/poster for presentation at a national conference, a manuscript for submission to a peer-reviewed journal).

NIS Protocol 

**Study number: 1199-0526 Document number: c41847952-01** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

- 1. Meltzer, EB, Noble, PW. Idiopathic pulmonary fibrosis. Orphanet journal of rare diseases. 2008; 3(1), 1-15.
- 2. Strongman H, Kausar I, Maher TM. Incidence, prevalence, and survival of patients with idiopathic pulmonary fibrosis in the UK. Adv Ther. 2018;35(5):724–36.
- 3. Raghu G, Rochwerg B, Zhang Y, Garcia CA, Azuma A, Behr J, et al; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT clinical practice guideline: treatment of idiopathic pulmonary fibrosis. An update of the 2011 clinical practice guideline, Am J Respir Crit Care Med 2015; 192: e3–19.
- 4. U.S. Food and Drug Administration. News release. FDA approves Esbriet to treat idiopathic pulmonary fibrosis. October 15, 2014. Available at: http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm418991.html
- 5. U.S. Food and Drug Administration. News release. FDA approves Esbriet to treat idiopathic pulmonary fibrosis. October 15, 2014. Available at: http://www.fda.gov/NewsEvents/Newsroom/PressAnnouncements/ucm418991.html
- 6. Paterniti MO, Bi Y, Rekić D, Wang Y, Karimi-Shah BA, Chowdhury BA. Acute exacerbation and decline in forced vital capacity are associated with increased mortality in idiopathic pulmonary fibrosis. Ann Am Thorac Soc. 2017;14(9):1395–402.
- 7. King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, et al.; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014; 370:2083–2092.
- 8. Richeldi L, du Bois RM, Raghu G, Azuma A, Brown KK, Costabel U, et al.; INPULSIS Trial Investigators. Efficacy and safety of nintedanib in idiopathic pulmonary fibrosis. N Engl J Med. 2014; 370:2071–82.
- 9. Dempsey T, Sangaralingham LR, Yao X, Sanghavi D, Shah ND, Limper AH. Clinical Effectiveness of Antifibrotic Medications for Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med 2019; Iss 2, pp 168–174
- 10. Corral M, Reddy S, Chang E, Broder M, Gokhale S, Raimundo K. Rates of Adherence and Persistence of Antifibrotic Therapies in the U.S. Medicare Population. Poster presented at: American Thoracic Society 2019 International Meeting; 2019 May 17–22; Dallas, TX.
- 11. Corral M, DeYoung K, Kong AM. Treatment patterns, healthcare resource utilization, and costs among patients with idiopathic pulmonary fibrosis treated with antifibrotic medications in US-based commercial and Medicare Supplemental claims databases: a retrospective cohort study. BMC Pulm Med. 2020 Jul 11;20(1):188. doi: 10.1186/s12890-020-01224-5.

NIS Protocol 
Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- 12. Nathan SD, Lancaster LH,2 Albera C, Glassberg MK, Swigris JJ, Gilberg F, et al.; Dose modification and dose intensity during treatment with pirfenidone: analysis of pooled data from three multinational phase III trials. BMJ Open Resp Res 2018;5:e000323. doi:10.1136/bmjresp-2018-000323
- 13. Genentech. https://www.gene.com/download/pdf/esbriet\_prescribing.pdf. Accessed 09/26/2022, 2022
- 14. PI BI. https://docs.boehringer-ingelheim.com/Prescribing%20Information/PIs/Ofev/ofev.pdf. Accessed 09/26/2022, 2022
- 15. Data on File, Boehringer Ingelheim, Nintedanib (BIBF 1120) Summary of Clinical Efficacy, Document Number: c02155681-02

NIS Protocol 

**Study number: 1199-0526 Document number: c41847952-01** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **ANNEXES**

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

| Number | Document<br>Reference<br>Number | Date | Title |
|--------|---------------------------------|------------|---------------------|
| 1 | <number></number> | 11/12/2021 | 1276_Code_List.xlsx |

NIS Protocol 

**Study number: 1199-0526 Document number: c41847952-01** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS



ENCePPChecklistforSt

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **ANNEX 3. ADDITIONAL INFORMATION**

Not applicable

NIS Protocol 

Study number: 1199-0526 Document number: c41847952-01

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES

The NIS Protocol must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global<br>NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi | X | X | X |
| Global TMM / TMMA / TM<br>Market Access | X | X | |
| Global Project Statistician | X | X | |
| Global TM RA | X | | |
| Global PVWG Chair | X | | |
| GPV SC | X | X | X |
| Global CTIS representative | X | | |
| Local Medical Director | X (if local study) | | X |
| Local Head MAcc / HEOR<br>Director | X (if local study) | | X |
| Global TA Head Epi* | X | X | |
| Global TA Head Clinical Development / Medical Affairs / Market Access* | X | X | |
| Global TA Head PV RM* | X | | |
| RWE CoE | X | X | |
| PSTAT / PSTAT-MA (for NISnd only) | X | X | X |
| NIS DM | X | X | X |
| Local Head MA/Clinical<br>Development | | | X (does not apply to<br>NISed without chart<br>abstraction) |

<sup>\*</sup> After review by Global TM for function

Include this Annex if signatures of external investigators are required **and/or** for studies that will not be stored in the DMS for submission documents. For non-interventional studies

NIS Protocol 

**Study number: 1199-0526 Document number: c41847952-01** 

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

approval signatures must be obtained from the individuals as noted in section 5.1.3 "Manage NIS Protocol" in the corresponding SOP 001-MCS-90-118. If the study is a PASS, additional approvals are necessary; refer to SOP 001-MCS-90-140 "Post Authorization Safety Studies".

| Study Title: | | |
|---|---|---|
| Study Number: | | |
| Protocol Version: | : | |
| I herewith certify referenced in the | that I agree to the content of the study study protocol. | protocol and to all documents |
| Note: Please insert | t respective signatories with regard to the | SOP. |
| Position:I_ | Name/Date: | y> Signature: |
| Position: NIS | Name/Date: ≤ / dd mmm yyyy | > Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |